CLINICAL TRIAL: NCT07067567
Title: A Phase Ia Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Anti-tumor Efficacy of AK146D1 for Injection, an Anti-Trop2/Nectin4 Bispecific Antibody-drug Conjugate, in Patients With Advanced Solid Tumors
Brief Title: A Study of AK146D1 for Injection in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AK146D1-101
Record Dates: First submitted 2025-06-18; First posted 2025-07-16 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AK146D1 for injection (Experimental): AK146D1 for injection will be administered in prespecified dose levels
  Interventions: Drug: AK146D1 for injection

INTERVENTIONS:
Drug: AK146D1 for injection — AK146D1 for injection is an anti-Trop2/Nectin4 bispecific antibody-drug conjugate

SUMMARY:
This is an first-in-human, Phase I clinical study aimed at evaluating the safety, tolerability, PK, immunogenicity, and preliminary antitumor efficacy of AK146D1 for injection in advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to understand and voluntarily sign the written informed consent form.
2. Aged of ≥ 18 years and ≤75 years.
3. ECOG PS 0 or 1.
4. The expected lifespan is ≥3 months.
5. Histologically-confirmed unresectable advanced solid tumors with disease progression or intolerance to standard treatment or no standard treatment available.
6. At least one measurable lesion according to RECIST v1.1.
7. Have sufficient organ function.
8. Females subjects must not be pregnant at screening or have evidence of non-childbearing potential. Agree to use medically accepted methods of contraception

Exclusion Criteria:

1. Having other active malignancies within 3 years.
2. Currently participating in another interventional clinical study.
3. Presence of active metastases to the central nervous system. For patients with asymptomatic brain metastasis or stable symptoms after treatment can be included.
4. Having received any treatment targeting Trop2 or Nectin4.
5. Having received systemic anti-tumor treatment within 4 weeks or 1 cycle interval of the regimen or major surgical operations within 4 weeks before the first administration.
6. Toxicity of previous antineoplastic therapy has not resolved to NCI CTCAE 5.0 grade 1 or lower.
7. Subjects with clinically significant cardiovascular or cerebrovascular diseases or risks.
8. Subjects with active autoimmune diseases requiring systemic treatment within 2 years.
9. Known active infection requiring antibodies treatment within 2 weeks, or severe infection within 4 weeks prior to the first dose.
10. Known to be positive for HIV and other infections.
11. Previous history of severe hypersensitivity reactions.
12. Live attenuated vaccines were received within 4 weeks.
13. Subjects with a history of mental illness and incapacitated or limited capacity.
14. Any disease or condition that, in the opinion of the investigator, would compromise subject safety or interfere with study assessments.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2026-11-05 (Estimated); Study Completion 2027-05-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities (DLTs) | During the first 3 weeks of treatment.
  DLTs are defined as toxicities that meet pre-defined severity criteria, and assessed as having a suspected relationship to study drug.
Number of participants with adverse events (AEs) | From the time of signing informed consent form through 30 days(for AEs) or 90 days(for SAEs) after the last dose of study drug.
  AEs refer to any untoward medical occurrence or deterioration of existing medical events after the participants sign the ICFs, whether or not considered related to the study treatment.

SECONDARY OUTCOMES:
Serum PK concentration of AK146D1 | From pre-dose to the end of the last dose, an average of 6 months.
  Serum PK concentration of AK146D1 in participants after administration
Anti-drug antibodies (ADA) | From pre-dose to 30 days post end of treatment
  The number and percentage of participants with detectable anti-drug antibodies (ADA)
Objective Response Rate (ORR) assessed by investigator per RECIST v1.1 | Up to approximately 2 years
  ORR is the proportion of participants with complete response(CR) or partial response(PR) , assessed based on RECIST v1.1.
Disease Control Rate (DCR) assessed per RECIST v1.1 | Up to approximately 2 years
  DCR is defined as the proportion of participants with CR, PR, or SD, assessed based on RECIST v1.1.
Duration of response (DoR) assessed by the investigator per RECIST v1.1 | Up to approximately 2 years
  DoR is defined as the duration from the first documentation of objective response to the first documented disease progression (based on RECIST Version 1.1) or death due to any cause, whichever occurs first.
Time to response (TTR) assessed by the investigator per RECIST v1.1 | Up to approximately 2 years
  TTR is defined as the time to objective response based on RECIST v1.1.
Progression Free Survival (PFS) assessed by investigator per RECIST v1.1 | Up to approximately 2 years
  PFS is defined as the time from the start of treatment until the first documentation of disease progression (based on RECIST Version 1.1) or death due to any cause, whichever occurs first.
Overall survival (OS) | Up to approximately 2 years
  OS is defined as the time from the first dose to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- SunYat-sen University Cancer Center, Guangzhou, Guangdong, China